CLINICAL TRIAL: NCT04080661
Title: Evaluation of the Predictive Value of Early Serum Trough Concentrations and Anti-drug Antibodies of Secukinumab and the Development of a Concentration Response Curve of Secukinumab for Psoriasis Patients.
Brief Title: Therapeutic Drug Monitoring of Secukinumab in Psoriasis Patients.
Acronym: BIOLOPTIM-SEC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: KU Leuven (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BC-02602 - BIOLOPTIM-SEC
Record Dates: First submitted 2019-07-19; First posted 2019-09-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Psoriasis Vulgaris
Keywords: Therapeutic drug monitoring; Psoriasis; Secukinumab
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: A prospective, open label, non-randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Standard of care - secukinumab (Experimental): Patients will continue to receive secukinumab according to the standard dosing schedule: subcutaneous injections once a week for 5 weeks, then every 4 weeks (300 mg).
  Interventions: Procedure: Venapuncture; Other: Patient questionnaires

INTERVENTIONS:
Procedure: Venapuncture — Blood samples will be collected to determine the serum trough levels and anti-drug antibodies of secukinumab.
Other: Patient questionnaires — The study participants will complete the Dermatology Quality of Life (DLQI) and EQ-5D-5L questionnaire at each study visit.

SUMMARY:
Biologics such as secukinumab are currently the most effective treatment option for patients with moderate to severe psoriasis. But they are costly for healthcare systems and still described according to a'one dose fits all' dosing regimen, leading to potential over-and undertreatment. In this study we aim to investigate the predictive value of early serum trough levels of secukinumab and determine the therapeutic window of secukinumab in psoriasis patients.

DETAILED DESCRIPTION:
Patients will be included after signing informed consent. After inclusion, patients will continue on standard dosing schedule of secukinumab (i.e. subcutaneous injections once a week for 5 weeks (300 mg) followed by subcutaneous injections every 4 weeks). During each study visit blood will be taken in order to quantify Ctroughs and/or anti-drug antibodies towards secukinumab. In addition, Psoriasis Area and Severity Index (PASI) and Investigator's Global Assessment (IGA) score will be evaluated by a physician. Patients complete the Dermatology Life Quality Index (DLQI) and European quality of life EQ-5D instrument at each visit.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have a clinical or histological diagnosis of chronic plaque-type psoriasis
2. Participants must sign an ICF indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study

Exclusion Criteria:

1. Participants who have currently a predominant nonplaque form of psoriasis
2. Participants who are pregnant, nursing or planning a pregnancy
3. Participants who are unable or unwilling to undergo multiple venapunctures
4. Participants who are treated according to a different dosing schedule than standard dosing of secukinumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive value of early serum trough concentrations of secukinumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 24 based on serum trough concentrations of secukinumab measurements taken from week 0,1,2,3 and/or 4.
Predictive value of early anti-drug antibodies of secukinumab | Week 0 until week 24 of treatment
  Prediction of the clinical response (PASI) at week 12 and/or week 24 based on anti-drug antibodies (ADA) measurements taken from week 0,1,2,3 and/or 4.
Development of the therapeutic window of secukinumab in psoriasis | Week 0 until week 52 of treatment
  Defining a therapeutic window for secukinumab based on serum trough concentrations corresponding with adequate clinical response

SECONDARY OUTCOMES:
DLQI | Week 0 until week 52 of treatment
  The DLQI (Dermatology Life Quality Index) (range 0-30) is a dermatology specific quality of life (QoL) instrument designed to assess the impact of the disease on participant's QoL. It is a ten item questionnaire that, in addition to evaluated overall QoL, can be used to assess six different aspects that may affect QoL: 1) symptoms and feelings, 2) daily activities, 3) leasure, 4) work or school performances, 5) personal relationships, and 6) treatment.
  The scoring of each question is as follows:
  Very much - scored 3; A lot - scored 2; A little - scored 1; Not at all - scored 0; Not relevant - scored 0; Question 7, 'prevented work or studying' - scored 3. The DLQI is calculated by summing the score of each question resulting in a maximum of 30 and a minimum of 0. The higher the score, the more quality of life is impaired.
EQ-5D-5L | Week 0 until week 52 of treatment
  The EQ-5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits of the five dimensions can be combined into a 5- digit number that describes the patients' health state.
EQ VAS | Week 0 until week 52 of treatment
  The EQ VAS (Visual Analogue Scale) (range 0-10) records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.

CONTACTS AND LOCATIONS:
Overall Officials: Jo Lambert, Prof., Principal Investigator — University Ghent
Locations (7):
- Belgium (7):
  - AZ Maria Middelares, Ghent, East-Flanders
  - AZ Sint-Lucas, Ghent, East-Flanders
  - University Hospital Ghent, Ghent, East-Flanders
  - Private practice Dermatology, Maldegem, East-Flanders
  - University Hospital Leuven, Leuven, Vlaams-Brabant
  - AZ Sint-Jan, Bruges, West-Flanders
  - AZ Delta Rembert, Torhout, West-Flanders

IPD SHARING:
Plan to Share IPD: No